CLINICAL TRIAL: NCT04070118
Title: Evaluation of Lower Uterine Segment Thickness in Pregnant Women Presenting With Term Pain and Previous Cesarean Section
Brief Title: Lower Uterine Segment Thickness and Term Pain,Previous Cesarean Section
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, pınar kadiroğulları M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.05.117
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cesarean Section; Dehiscence; Cesarean Section Complications
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with previous cesarean section: presenting to the emergency department with pain, previous cesarean section; Patients measured niche thickness before operation
  Interventions: Procedure: Measure niche thickness with ultrasound

INTERVENTIONS:
Procedure: Measure niche thickness with ultrasound — in patients with previous cesarean section who applied to the emergency department with pain and underwent surgery; Measure niche thickness before operation

SUMMARY:
the purpose of the researchers; The aim of this study is to evaluate the consistency of niche dimensions measured by ultrasonography with visual measurement of the surgeon during the operation of the patient when presenting with pain in her current pregnancy.

If patients who have had previous cesarean section present to the emergency department with pain or NST pain, a panic occurs immediately for operation. Purpose of researchers; The aim of this study is to investigate whether a really fine determination of the thickness of the old incision line is associated with full-thickness rupture or incomplete rupture, which appears to be an operation, and if a relationship is found, there is a limit for this thickness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous cesarean section
* Those in term gestational week (37-42 weeks)
* Those who apply to the emergency with pain

Exclusion Criteria:

* Birden fazla sezaryen geçirilmiş öyküsü olan hastalar
* Önceden geçirilmiş uterin cerrahisi olan hastalar
* Miad olmayan gebeler
* Plesantal yerleşim patolojısı olan gebeler

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In Pregnant Women with Term Pain and Previous Cesarean Section; Patients with visual evaluation of the lower uterine segment thickness and ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Measure niche thickness with ultrasound | 1 day
  Ultrasonography of Lower Uterine Segment Thickness in Pregnant Women Presenting with Term Pain and Previous Cesarean Section It will be given in mm.
Measure niche thickness with visual evaluation of the surgeon | 1 day
  Measured Lower Uterine Segment Thickness by Visual Evaluation of Pregnant Women Presenting with Term Pain and Previous Cesarean Section no rupture have full coat rupture have incomplete rupture; will be valued as.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)